CLINICAL TRIAL: NCT04430309
Title: The Feasibility and Efficacy of Baduanjin Exercise on Cognition and Physical Fitness Among Patients With Schizophrenia:Randomized Controlled Trial
Brief Title: Baduanjin on Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Taiwan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202000817B0
Record Dates: First submitted 2020-06-03; First posted 2020-06-12 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia
Keywords: Schizophrenia, mind body intervention ,Baduanjin
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Baduanjin exercise group (Experimental): The intervention group will practice Badunjin in a group which include 6-8 participants and one trained medical staff. The Baduanjin is an ancient Chinese mind-body exercise, which comprised of eight simple movements.
  The sessions will take place twice a week, 60 minutes per session for a total duration of 12 weeks
  Interventions: Behavioral: Baduanjin exercise program
- Control group (Active Comparator): The control group will receive brisk walking activities. The sessions will take place twice a week, 60 minutes per session for a total duration of 12 weeks
  Interventions: Behavioral: Brisk walking program

INTERVENTIONS:
Behavioral: Baduanjin exercise program — The sessions includes 10-minute warm-up, 40-minute Baduanjin exercise and 10-minute cool down.
  Other Names: Eight Silken Movements; Eight Silk Weaving
  Arms: Baduanjin exercise group
Behavioral: Brisk walking program — The sessions includes 10-minute warm-up, 40-minute brisk walking and 10-minute cool down.
  Arms: Control group

SUMMARY:
As an ancient, popular Chinese exercise, Baduanjin is characterized by symmetrical posture, deep breathing and meditation and easy to learn. Previous studies showed immediate effect of Baduanjin on cognition in patients with schizophrenia.The purpose of this study is to investigate the immediate effect and chronic effect of Baduanjin exercise on physical fitness, cognition and daily functions in middle-aged and older adults with schizophrenia.

DETAILED DESCRIPTION:
A single-blind, 2-arm randomized controlled trial investigating the benefits of Baduanjin exercise on middle-aged and older patients with schizophrenia. A total of 48 participants will be assigned to either 12 weeks of 60-minute two sessions per week Baduanjin exercise group or a brisk walking group. Primary outcomes are physical fitness and cognition functions. Secondary outcomes are dual task performance and daily functions. Evaluation will be completed at baseline, immediately after treatment and 4-week follow up.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of schizophrenia according to the DSM-5.
* Independent adult aged 40 years or older in the day-care center.
* Having a stable mental status without shift in medication and keep in same dose for at least one month.

Exclusion Criteria:

* Serious physical conditions that will impede participation, such as cardiovascular disease, musculoskeletal disease or pulmonary system disease.
* Visual or auditory impairment that precludes completion of assessment.
* Acute psychosis requiring hospitalization.
* Presence of severe withdrawal or profound cognitive disability that cause difficulties in following instructions.
* Participating in another clinical trial at the same time.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change scores of 6-minute walk test | Baseline, immediate after treatment, 4-week follow up
  This test evaluates cardiovascular fitness and walking speed.
Change scores of 30-second chair stand test | Baseline, immediate after treatment, 4-week follow up
  This test evaluates muscular endurance of lower-extremities.
Change scores of Timed up-and-go test | Baseline, immediate after treatment, 4-week follow up
  This test evaluates functional mobility, agility and balance
Change scores of Montreal cognitive assessment | Baseline, immediate after treatment, 4-week follow up
  This test evaluates global cognition.
Change scores of Trail making test (part A and part B) | Baseline, immediate after treatment, 4-week follow up
  This test evaluates speed of processing, visual attention and cognitive flexibility.
Change scores of Logical Memory | Baseline, immediate after treatment, 4-week follow up
  It is a subtest of the Wechsler Memory Scale. This test evaluates memory.

SECONDARY OUTCOMES:
Change scores of dual task Timed up-and-go test (manual) | Baseline, immediate after treatment, 4-week follow up
  This test requires carry a cup of water 3 cm from the top of the cup while performing the Timed up-and-go test. It evaluates dual task performance.
Change scores of dual task Timed up-and-go test (cognitive) | Baseline, immediate after treatment, 4-week follow up
  This test combine serial three counting and Timed up-and-go test simultaneously. It evaluates dual task performance.
Change scores of Activities of Daily Living Rating Scale III | Baseline, immediate after treatment, 4-week follow up
  It is a self-administered, paper-and-pencil test that evaluates daily functions

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung Medical Center, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided